CLINICAL TRIAL: NCT06386276
Title: Surgical TReatment of Women With Deep ENDometriosis Infiltrating the Sigmoid Colon and/or the Rectum. A Monocentric Archive
Brief Title: Surgical TReatment of Women With Deep ENDometriosis
Acronym: TrEnd
Status: Recruiting | Type: Observational
Sponsor: Casa di Cura Privata 'Malzoni - Villa dei Platani' S.P.A. (Other)
Responsible Party: Principal Investigator, Francesca Falcone, Medical Doctor, Casa di Cura Privata 'Malzoni - Villa dei Platani' S.P.A.
Other Study IDs: 00025986
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Deep Endometriosis; Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colorectal bowel resection — The TrEnd is a single-institutional retrospective/prospective study, conducted in a high-volume referral centre for the endometriosis diagnosis and management, with the aim of systematically collecting data from consecutive patients undergoing segmental sigmoid colon/rectal resection for deep endometriosis.

SUMMARY:
TrEnd trial is aimed to collect data from consecutive patients undergoing segmental sigmoid colon/rectal resection for deep endometriosis. The main purpose of this project is to gather a large series of cases treated using standardized surgical procedures, allowing a precise evaluation of complications and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 18 years;
* presence of deep endometriotic nodule(s) infiltrating the tunica muscularis of the sigmoid colon/rectum.

Exclusion Criteria:

* age <18 years:
* presence of coexisting inflammatory bowel disease;
* patients who have received previous pelvic radiotherapy.

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women undergoing segmental sigmoid colon/rectal resection for deep endometriotic nodules infiltrating the tunica muscularis of the sigmoid colon/rectum preoperatively identified with imaging and surgically treated with segmental resection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
To document the surgical strategies adopted for treating patients with deep endometriosis undergoing to sigmoid colon/rectal resection | 10 years
  Percentage
To assess the rate of complications | 10 years
  Rate/percentage
To assess the rate of conversion to open surgery | 10 years
  Rate/percentage
To assess the rate of endometriosis-free bowel resection margins | 10 years
  Rate/percentage
To assess the rate of recurrence | 10 years
  Rate/percentage

SECONDARY OUTCOMES:
To assess the intraoperative blood loss | 10 years
  Median with IQR
To assess the operating time | 10 years
  Median time with IQR
To assess the gastrointestinal function recovery | 10 years
  Median days with IQR
To assess the duration of hospital stay | 10 years
  Median days with IQR
To assess the reproductive outcomes | 10 years
  Rate/percentage of pregnancies, normal full term deliveries, spontaneous and voluntary abortions

CONTACTS AND LOCATIONS:
Overall Officials: Mario Malzoni, MD, Principal Investigator — malzonimario@gmail.com; Francesca Falcone, MD, Principal Investigator — francescafalcone@malzoni.org
Locations (1):
- Casa Di Cura Malzoni Villa Platani Spa, Avellino, Campania, Italy

IPD SHARING:
Plan to Share IPD: Undecided